CLINICAL TRIAL: NCT03063554
Title: Endoscopic Ultrasound-Guided Biliary Drainage (EUS-BD) Compared to Standard Transpapillary Biliary Drainage (ERCP-TP) for Palliation of Jaundice in Unresectable Cancer of the Head of the Pancreas (BILPAL TRIAL)
Brief Title: EUS BD vs ERCP TP for Pancreatic Cancer
Acronym: BILPAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief of Endoscopy, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1603017104
Record Dates: First submitted 2017-02-16; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer; Pancreatic Adenocarcinoma; Biliary Tract Neoplasms; Biliary Duct Obstruction; Unresectable Pancreatic Cancer; Periampullary Cancer; Periampullary Carcinoma Non-Resectable
Keywords: Endoscopy; Pancreatic Cancer; Bile duct; Periampullary; ERCP; Biliary drainage; Biliary obstruction; EUSBD; TEUS; EUS; Endoscopic Ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Ultrasound Guided Biliary Drainage (Active Comparator): Endoscopic Ultrasound Guided biliary drainage with stent placement. EUS via either stomach or duodenum.
  Interventions: Procedure: Endoscopic Ultrasound Guided Biliary Drainage
- ERCP (Placebo Comparator): Endoscopic Retrograde Cholangiopancreatography with transpapillary biliary stent placement only.
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: Endoscopic Ultrasound Guided Biliary Drainage — Endoscopic Ultrasound Guided biliary drainage with stent placement;
  Other Names: EUSBD
  Arms: Endoscopic Ultrasound Guided Biliary Drainage
Procedure: ERCP — Endoscopic Retrograde Cholangiopancreatography with transpapillary biliary stent placement
  Other Names: ERCP-TP
  Arms: ERCP

SUMMARY:
This Endoscopic Ultrasound guided Biliary Drainage (EUS-BD) vs. Endoscopic Retrograde Cholangiopancreatography (ERCP-TP) trial (BILPAL) is a randomized controlled multicenter trial that will provide evidence whether or not traditional ERCP biliary drainage is to be performed in patients with obstruction in bile duct due to unresectable pancreatic head or periampullary tumor.

DETAILED DESCRIPTION:
Obstructive jaundice is the most common symptom in patients with periampullary cancer and cancer of the pancreatic head. For patients with unresectable tumors, palliation of malignant obstructive is traditionally achieved using endoscopic retrograde cholangiopancreatography (ERCP) with transpapillary (TP) stent placement. Data show that ERCP is equivalent to surgery with regards to relief of jaundice. Self-expandable metal stents (SEMS) offer prolonged palliation compared to large-bore (10Fr) plastic stents. However, it is believed that gastric outlet obstruction occurs more commonly in patients who have received SEMS for palliation of MOJ. In addition, ERCP is associated with adverse events including pancreatitis, post-sphincterotomy bleeding, and perforation.

More recently endoscopic ultrasound (EUS)-guided biliary drainage has been described for biliary drainage in patients with malignant distal bile duct obstruction. Thus far it has been used as a rescue approach when traditional ERCP-guided transpapillary biliary drainage ERCP fails. TP failure can occur as a result of duodenal obstruction, failed cannulation, and failed wire access across the stricture.

Potential advantages of EUS-guided biliary drainage include avoidance of pancreatitis and post-sphincterotomy bleeding. Additionally, it may result in a lower frequency of gastric outlet obstruction since the stent does not encroach upon the tumor.

To compare the potential advantages of EUS-guided biliary drainage the investigators are conducting a multicenter, randomized trial comparing the EUS-guided drainage to traditional ERCP.

This EUS-BD vs. ERCP-TP-trial (BILPAL) is a randomized controlled multicenter trial that will provide evidence whether or not traditional ERCP biliary drainage is to be performed in patients with obstruction in bile duct due to unresectable pancreatic head or periampullary tumor.

This study will enroll 120 subjects; 60 subjects in each arm. Trial duration is about 1 year and involves 5-7 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 90 years old
2. Clinically indicated for biliary endoscopic drainage with Endoscopic Ultrasound guidance or ERCP
3. CT scan has demonstrated a lesion in the pancreatic head area with metastases and/ or local tumor ingrowth preventing resection.
4. CT with evidence of distant metastases or local tumor ingrowth into portal or mesenteric vessels (as defined by the tumor surrounding the vessel for at least 180 degrees of the circumference)
5. A serum bilirubin level of > 2.5mg/dL at randomization
6. Deemed surgically unresectable
7. Consents to participation in the randomized controlled trial

Exclusion Criteria :

1. > 90 years
2. Severe comorbidity (Karnofsky <50%)
3. Any prior successful previous biliary drainage including ERCP and stenting, percutaneous biliary and surgical,
4. Prior surgically altered pancreaticobiliary or gastroduodenal anatomy.
5. Female of childbearing potential with a positive pregnancy test prior to the procedure or intends to become pregnant during the study.
6. Currently participating in another device trial that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10-18 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Stent Patency | 6 months after randomization
  Efficacy is measure by the evaluation of biliary stent patency at month 6 post randomization

SECONDARY OUTCOMES:
Safety evaluation: Assessment of number and frequency of procedure related adverse events within 1 month of the procedure | Within 1 month of procedure
  Assessment of number and frequency of procedure related adverse events within 1 month of the procedure
Clinical Success | 1 month from procedure
  Resolution of jaundice due to obstruction in the bile duct
Technical Success | 1 month from procedure
  Technical success is defined as successful stent insertion providing biliary drainage with confirmation of appropriate radiographic positioning
Survival duration | 2 years from randomization
  Survival duration will be measured from time of diagnosis to death
Serum bilirubin decrease | 1 month from procedure
  Duration to achieving at least 30% decrease in serum bilirubin or normalization of serum bilirubin level (≤1.2 mg/dL)
Quality of Life | 1 year from study enrollment
  QOL will be measured via QLQ-C30 questionnaires completed by the subject at each follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No